CLINICAL TRIAL: NCT00277381
Title: Improving Adherence in Patients With Hypertension - A Novel Use of Communication Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Director, Center for Connected Health, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 2005-P-002248
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Hypertension
Keywords: Adherence; Hypertension; Telemedicine
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Automated feedback regarding drug adherence

SUMMARY:
Treating hypertension is known to decrease morbidity and mortality. Despite this 70% of patients do not have adequately controlled blood pressure. The main reason for this is non-adherence to recommended drug therapy. Although strategies have been developed to improve adherence many are time consuming and expensive. We propose to use communications technology to develop a novel means of improving adherence to antihypertensive therapy. We will conduct a randomised, single-blinded, controlled study to assess the impact of a real-time, automated reminder system on adherence rates. This will involve adapting two pieces of currently available technology - the electronic pill bottle and the Ambient Globe. The Globe will change colour in response to information received, via a wireless link, from the patient's electronic pill bottle. We hypothesise that this will provide patients with an up to date, but unobtrusive, reminder of their adherence status and thus effect positive behavioural change. We will measure the impact of this intervention on adherence rates as well as assessing patient views and the impact on provider workload. This trial will elucidate the role of communications technology in improving adherence behaviour and allow us to develop further strategies to tackle this major health issue.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of a once-a-day dose of atenolol.
* Morisky Score of less than or equal to 2 (explanation in 'Equitable Selection of Subjects').
* Fluency in English.
* Age 45-65 inclusive.
* Primary Care Physician consent to the patient taking part.

Exclusion Criteria:

* Patients prescribed more than two anti-hypertensive agents.
* Patients prescribed more than four medications in total.
* Patients on secondary prevention following cardiac event or stroke.
* Morisky Score of more than 2.
* Patients with visual impairment or color-blindness.
* Patients with congenital or acquired cognitive impairment.
* Patients with a cardiac pacemaker

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Adherence rates as measured using data held in the SIMpill database
Patient satisfaction with intervention as assessed by questionnaire at the end of the study.
Technical difficulties as assessed by interview at the end of the study and by review of the technical log.

SECONDARY OUTCOMES:
Discontinuation rates of medication as assessed at the end of trial debrief.
Changes to medication regime as assessed at the end of trial debrief.
Adverse events (e.g. hospitalisation) as assessed from the log of withdrawals from the trial.
Blood pressure as measured on enrollment and at end of trial debrief.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Kvedar, MD, Principal Investigator — Partners Healthcare System
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States